CLINICAL TRIAL: NCT01059357
Title: A Pilot Study Assessing Transoral Robotic Surgery (TORS) for Oral and Laryngopharyngeal Benign and Malignant Lesions Using the Da Vinci Robotic Surgical System
Brief Title: Transoral Robotic Surgery (TORS) for Oral and Laryngopharyngeal Lesions Using Da Vinci Robotic Surgical System
Acronym: TORS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00009802; CCCWFU 60209 (Other: Wake Forest University Health Sciences)
Record Dates: First submitted 2010-01-21; First posted 2010-01-29 (Estimated); Results first posted 2018-11-16 (Actual); Last update posted 2018-11-16 (Actual); Status verified 2018-11

CONDITIONS: Head and Neck Neoplasms
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Transoral Robotic Surgery (TORS) (Experimental): Transoral Robotic Surgery (TORS) using the Da Vinci Robotic Surgical System
  Interventions: Device: Da Vinci Robotic Transoral Robotic Surgical System

INTERVENTIONS:
Device: Da Vinci Robotic Transoral Robotic Surgical System — (TORS) Da Vinci Robotic Transoral Robotic Surgical System
  Other Names: (TORS) Da Vinci Robotic Transoral Robotic Surgical System

SUMMARY:
The purpose of this study is to conduct a pilot single-arm to assess transoral robotic surgery (TORS) for oral and laryngopharyngeal benign and malignant lesions using the Da Vinci Robotic Surgical System.

DETAILED DESCRIPTION:
Patients are going to be evaluated in their usual regular clinical follow ups starting with preoperative first visit, 3 weeks, 3 months and 6 months postoperatively with a Quality of Life survey (Head and Neck Cancer Inventory, HNCI-QOLQ).

ELIGIBILITY:
Inclusion Criteria:

* Patient must present with indications for diagnostic or therapeutic approaches for benign and malignant diseases of the oral cavity or laryngopharynx (including the neoplastic lesions of the tongue, tongue base, retromolar trigone, tonsils, palate, posterior and lateral pharynx, glottic, supraglottic and subglottic larynx)
* Patients must have adequate transoral exposure of the oral cavity and laryngopharynx for TORS instrumentation

Exclusion Criteria:

* Unexplained fever and/or untreated, active infection
* Patient pregnancy
* Previous head and neck surgery precluding transoral/robotic procedures
* The presence of medical conditions contraindicating general anesthesia or transoral surgical approaches

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2010-06 (Actual); Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joshua D. Waltonen, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Transoral Robotic Surgery (TORS)
Started | 58
Completed | 54
Not Completed | 4

BASELINE CHARACTERISTICS:
Arm/Group | Transoral Robotic Surgery (TORS)
Number analyzed (Participants) | 58
Age, Continuous [Mean (Full Range); unit: years] | 51.64 [27 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 43

OUTCOME MEASURES:

1. Primary Outcome: The Number and Percent of All Evaluable Patients Who Have Successfully Undergone TORS at Each Interim Analysis.
Description: In order to evaluate the feasibility of TORS, the investigators will report the number and percent of all evaluable patients who have successfully undergone TORS at each interim analysis
Time Frame: At time of surgery, lasting up to 3 hours. Assessed for up to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Transoral Robotic Surgery (TORS)
Number analyzed (Participants) | 58
Participants | 54

2. Secondary Outcome: Operative Time
Description: The total operative times include the induction of and emergence from anesthesia, the TORS procedure, plus any adjunct procedures (eg, neck dissections) performed during the same operation.
Time Frame: At time of surgery, up to 3 hours
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Transoral Robotic Surgery (TORS)
Number analyzed (Participants) | 54
minutes | 321 (136.63)

3. Secondary Outcome: Number of Participants With Blood Loss and Complications
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Transoral Robotic Surgery (TORS)
Number analyzed (Participants) | 54
Participants | 7

4. Secondary Outcome: Average Time to Set up and Perform Procedures
Description: This outcome is to identify the learning curve for TORS by measuring the efficiency of the surgeon who performs the procedures.
Time Frame: At time of surgery, up to 3 hours
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Transoral Robotic Surgery (TORS)
Number analyzed (Participants) | 54
minutes | 109 (47.1)

5. Secondary Outcome: Number of Correctly Predicted Success of TORS Preoperatively
Description: This outcome is to identify the learning curve for TORS by measuring the accuracy of the surgeon who performs the procedures.
Time Frame: preoperative
Measure: Number; unit: procedures
Arm/Group | Transoral Robotic Surgery (TORS)
Number analyzed (Participants) | 54
procedures | 53

6. Secondary Outcome: QOL
Description: Quality of life (QOL) of the patients undergoing TORS will be measures. The score range is 0-100 with higher scores denoting better outcome.
Time Frame: 6 months
Population: Data not collected on all participants
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Transoral Robotic Surgery (TORS)
Number analyzed (Participants) | 42
score on a scale | 52 (13.2)

ADVERSE EVENTS:
Time Frame: up to 6 months
Arm/Group | Transoral Robotic Surgery (TORS)
All-Cause Mortality (participants affected / at risk) | 0/54
Serious Adverse Events (participants affected / at risk) | 0/54
Other Adverse Events (participants affected / at risk) | 7/54
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Transoral Robotic Surgery (TORS) (N=54)
Blood loss (Blood and lymphatic system disorders) | 2
Chipped tooth (General disorders) | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1
Postoperative bleeding (Blood and lymphatic system disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes